CLINICAL TRIAL: NCT03532126
Title: A Prospective, Multi-center, Non-comparative, 52-week Follow-up, Post-market Clinical Investigation of Princess® VOLUME PLUS Lidocaine in Subjects With Midface Volume Deficit
Brief Title: A 52-week Clinical Investigation of Princess® VOLUME PLUS Lidocaine in Subjects With Midface Volume Deficit
Acronym: PRIMAvera
Status: Completed | Type: Observational
Sponsor: Croma-Pharma GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CPH-401-201331
Record Dates: First submitted 2018-04-24; First posted 2018-05-22 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Midface Volume Deficit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dermal filler for midface deficit: There will be one group in this study, the actual treatment group.
  Interventions: Device: Dermal filler for midface deficit

INTERVENTIONS:
Device: Dermal filler for midface deficit — During this procedure the device (a dermal filler) will be deep intradermal, subcutaneous or supraperiosteal injected according to its CE mark.

SUMMARY:
This investigation aims to confirm the safety and effectiveness of Princess VOLUME PLUS Lidocaine in midface volume deficit augmentation and includes a long term safety followup.

DETAILED DESCRIPTION:
This non-interventional study will evaluate subjects treated with Princess VOLUME PLUS Lidocaine for midface volume deficit augmentation. A touch-up treatment will be allowed, on discretion of the treating investigator, if the initial treatment didn't provide optimal correction. The effectiveness parameters will be evaluated based on a validated scale for midface volume deficit scale and confirmed by use of patient reported outcome questionnaires as well as based on photographs to be evaluated by an independent evaluator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older;
2. Presence of bilateral, approximately symmetric moderate to severe midface volume deficit, corresponding to MVDSS grades 2-3;
3. A negative urine pregnancy test at Visit 1 and commitment to use an adequate method of birth control for the duration of the clinical investigation (for women of childbearing potential only);
4. Healthy skin in the midface area and free of diseases that could interfere with evaluation of cutaneous aging or represent a risk for injection;
5. Willingness to abstain from any other aesthetic or surgical procedures in the treatment area for the duration of the investigation, including botulinum toxin injections (except glabella or forehead botulinum toxin treatment);
6. Capable to understand information about the investigation, including subjects' obligations, and is willing to take part, as evidenced by signed and dated informed consent.

Exclusion Criteria:

1. Presence or history of hypertrophic scarring, pigment disorders or keloid formation.
2. Presence or history of any autoimmune disease or current treatment with immune therapy.
3. History of hypersensitivity to hyaluronic acid, lidocaine hydrochloride or other amide-type local anaesthetics.
4. Previous treatment with a permanent filler in the area to be treated.
5. Pregnant or breastfeeding women.
6. Treatment with anticoagulants and platelet aggregation inhibitors (e.g., acetylsalicylic acid) within 10 days prior to Visit 1, unless the risk of bleeding/bruising is discharged after consultation with subject's physician who had prescribed such medicine.
7. Cutaneous, inflammatory and/or infectious processes (e.g., acne, herpes) in the area to be treated.
8. Laser therapy, dermabrasion or mesotherapy within 12 months, or chemical peeling within 3 months prior to Visit 1.
9. History of other aesthetic/surgical treatment which may interfere with performance evaluation.
10. Current or previous (within 30 days of enrolment) treatment with another investigational drug and/or medical device or participation in another clinical study.
11. Previous enrolment in this clinical investigation.
12. Any person dependent on the investigator (e.g., employees, relatives, or similar), or employees of the investigation site institution or the Sponsor.
13. The following subjects shall not participate: persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants (for Austria this is specified in the Medical Devices Act).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects suffering from moderate to severe midface volume deficit and having healthy skin in the treatment area.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Primary performance endpoint | 4 weeks
  Response rate at week 4 based on investigator's midface volume deficit severity scale (MVDSS) assessment, where response is defined as a MVDSS grade improvement by ≥1 grade compared to baseline.

SECONDARY OUTCOMES:
Secondary performance endpoint 1 | 12, 24, 36 and 52 weeks
  Response rate based on investigator's midface volume deficit severity scale (MVDSS) assessment.
Secondary performance endpoint 2 | 4, 12, 24, 36 and 52 weeks
  Global aesthetic improvement scale (GAIS) grade determined by the investigator.
Secondary performance endpoint 3 | 4, 12, 24, 36 and 52 weeks
  Global aesthetic improvement scale (GAIS) grade determined by the subject.
Secondary performance endpoint 4 | 4, 12, 24, 36 and 52 weeks
  Subject satisfaction.
Secondary performance endpoint 5 | 4, 12, 24, 36 and 52 weeks
  Response rate, based on midface volume deficit severity scale (MVDSS) assessment by the independent photography reviewer.
Secondary performance endpoint 6 | 4, 12, 24, 36 and 52 weeks
  Proportion of subjects with a midface volume deficit severity scale (MVDSS) grade improvement by ≥2 grades.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Prinz, Mag., Study Director — Sponsor GmbH
Locations (4):
- Austria (2):
  - Medizinisch Ästhetisches Zentrum Wien, Vienna
  - Yuvell, Vienna
- Germany (2):
  - Rosenpark Research, Darmstadt, Hesse
  - RZANY & HUND, Privatpraxis, Berlin

IPD SHARING:
Plan to Share IPD: No